CLINICAL TRIAL: NCT02657694
Title: Reviewing DAA Efficacy Managing Patient Treatment In Online Neighbourhoods
Acronym: REDEMPTION
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: FixHepC (Other)
Responsible Party: Sponsor
Other Study IDs: REDEMPTION
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination; Drugs, Generic; Sofosbuvir; daclatasvir; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Sofosbuvir+Ledipasvir: Following patients treating with Sofosbuvir+Ledipasvir
  Interventions: Drug: Sofosbuvir+Ledipasvir
- Sofosbuvir+Daclatasvir: Following patients treating with Sofosbuvir+Daclatasvir
  Interventions: Drug: Sofosbuvir+Daclatasvir
- Sofosbuvir+Velpatasvir: Following patients treating with Sofosbuvir+Velpatasvir
  Interventions: Drug: Sofosbuvir+Velpatasvir

INTERVENTIONS:
Drug: Sofosbuvir+Ledipasvir — DAA medication treatment
  Other Names: Harvoni (generic)
  Groups: Sofosbuvir+Ledipasvir
Drug: Sofosbuvir+Daclatasvir — DAA medication treatment
  Other Names: Sovaldi (generic); Daklinza (generic)
  Groups: Sofosbuvir+Daclatasvir
Drug: Sofosbuvir+Velpatasvir — DAA medication treatment
  Other Names: Epclusa (generic)
  Groups: Sofosbuvir+Velpatasvir

SUMMARY:
REDEMPTION (Reviewing DAA Efficacy Managing Patient Treatment In Online Neighbourhoods) is observing and collating the treatment course, safety profile, and outcomes of patients around the world who are choosing to self import generic versions of the Direct Acting Antivirals Sofosbuvir, Ledipasvir and Daclatasvir from countries like China, India and Bangladesh.

DETAILED DESCRIPTION:
The high prices of Hepatitis C Virus (HCV) Direct Acting Antiviral (DAA) medications in many countries have led patients to seek out less expensive generic alternatives.

The efficacy and safety of these generic medications has not been formally demonstrated in clinical practice.

The primary goal of REDEMPTION is to collate the clinical results of these generic medications.

The secondary goal is to answer efficacy questions for which there is currently insufficient trial data available - for example Sofosbuvir+Daclatasvir appears to be an inexpensive pan genotypic solution to treat HCV globally but this is supported by a total n of less than 1000, and in some common genotypes, such as HCV Genotype 2, by an n of only 52 making for a wide margin of error and a high degree of uncertainty.

ELIGIBILITY:
Inclusion Criteria:

Quantitative HCV RNA > 100

Exclusion Criteria:

Contraindications to DAA medications

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Worldwide, Hepatitis C Genotypes 1-6
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Sustained Virological Response 4 (SVR4) by Hepatitis C Virus (HVC) RNA Polymerase Chain Reaction (PCR) | 4-7 months
  Viral load 4 weeks after cessation of treatment as measured by HCV RNA PCR, where SVR is defined as HCV RNA < Lower Limit Of Quantification (LLOQ)

SECONDARY OUTCOMES:
Side Effects | 3-6 months
  Collating common side effects on treatment
Rapid Virological Response (RVR) by HCV RNA PCR | 4 weeks
  Viral load 4 weeks after starting treatment as measured by HCV RNA PCR
End Of Treatment (EOT) Response by HCV RNA PCR | 3-6 months
  Viral load at end of treatment as measured by HCV RNA PCR
Sustained Virological Response (SVR12) by HCV RNA PCR | 6-12 months
  Viral load 12 weeks after cessation of treatment as measured by HCV RNA PCR, where SVR is defined as HCV RNA < Lower Limit Of Quantification (LLOQ)

CONTACTS AND LOCATIONS:
Overall Officials: James Freeman, MB,BS,BSc, Study Director — ACRRM
Locations (1):
- FixHepC, Hobart, Tasmania, Australia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: REDEMPTION Website — http://fixhepc.com